CLINICAL TRIAL: NCT05027074
Title: A Randomized Parallel-group, Placebo-controlled, Double-blind, Event-driven, Multi-center Phase 2 Clinical Outcome Trial of Prevention of Arteriovenous Graft Thrombosis and Safety of MK-2060 in Patients With End Stage Renal Disease Receiving Hemodialysis
Brief Title: Global Study of MK-2060 (Anti-Factor XI Monoclonal Antibody) in Participants With End Stage Renal Disease Receiving Hemodialysis (FXI Hemodialysis Study) (MK-2060-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2060-007; MK-2060-007 (Other: MSD); 2024-511055-17-00 (Registry Identifier: EU CT); U1111-1303-0286 (Registry Identifier: UTN); 2020-002397-27 (EudraCT Number)
Record Dates: First submitted 2021-08-26; First posted 2021-08-30 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: End-Stage Renal Disease; End-Stage Kidney Disease; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-2060 20 mg (Experimental): MK-2060 20 mg administered via IV infusion during dialysis as a loading dose: QOD during week 1 (3 administrations), then QW after week 1
  Interventions: Drug: MK-2060
- MK-2060 6 mg (Experimental): MK-2060 6 mg administered via intravenous (IV) infusion during dialysis as a loading dose: Every other day (QOD) during week 1 (3 administrations), then once a week (QW) after week 1
  Interventions: Drug: MK-2060
- Placebo (Placebo Comparator): Placebo (normal saline) administered via IV infusion during dialysis as a loading dose: QOD during week 1 (3 administrations), then once a week after week 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-2060 — MK-2060 lyophilized powder diluted in normal saline and administered via IV infusion
  Arms: MK-2060 20 mg; MK-2060 6 mg
Drug: Placebo — Normal saline administered via IV infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two different doses of MK-2060 (a monoclonal antibody against Factor XI) in end stage renal disease (ESRD) participants receiving hemodialysis via an arteriovenous graft (AVG). Data from this study will be used to aid dose selection of MK-2060 in future studies. The primary hypothesis is that at least one of the MK-2060 doses is superior to placebo in increasing the time to first occurrence of AVG event.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of ESRD.
* Receiving hemodialysis (including hemodiafiltration) ≥3 times per week for a minimum of 3 hours per session via a mature normally functioning, uninfected AVG with at least 75% of the sessions meeting these criteria over the 4 weeks prior to randomization.
* A female participant is not pregnant or breastfeeding, not a woman of child-bearing potential (WOCBP) or is a WOCBP and agrees to follow contraceptive guidance during the intervention period and for at least 90 days after the last dose of study intervention.

Exclusion Criteria:

* Recent history of cancer (<1 year). Non-melanoma skin cancers are allowed.
* Mechanical/prosthetic heart valve.
* Recent hemorrhagic stroke or lacunar stroke (<1 month).
* Recent evidence (<1 month) of bleeding requiring hospitalization or unplanned medical attention, a history (≤2 years) of recurrent bleeding episodes including epistaxis, gastrointestinal (GI) bleeds or genitourinary (GU) bleeds requiring medical treatment or events requiring treatment with blood products.
* Recent history (<1 year) of drug or alcohol abuse or dependence.
* Currently receiving or planning to receive anticoagulants or antiplatelet medications (intradialytic heparin and aspirin are permitted).
* Planning on receiving a living donor renal transplant within 12 months (participants are permitted to be candidates for deceased donor renal transplants).
* Planning on receiving an arteriovenous fistula (AVF) placement within 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (120):
- United States (77):
  - Nephrology Consultants ( Site 0681), Huntsville, Alabama
  - AKDHC MEDICAL RESEARCH SERVICES, LLC-Maryvale ( Site 0723), Phoenix, Arizona
  - AKDHC Medical Research Services, LLC ( Site 0629), Tucson, Arizona
  - DaVita Anaheim West Dialysis-Davita Anaheim West Dialysis - Ismail ( Site 0562), Anaheim, California
  - DaVita Bakersfield Oak Street Dialysis-Clinical Research ( Site 0547), Bakersfield, California
  - Fresenius Kidney Care Bakersfield Northeast ( Site 0647), Bakersfield, California
  - Fresenius Kidney Care Meadows Field ( Site 0618), Bakersfield, California
  - California Institute Of Renal Research ( Site 0660), Chula Vista, California
  - Citrus Dialysis Center ( Site 0609), Covina, California
  - California Institute Of Renal Research ( Site 0679), El Centro, California
  - California Institute of Renal Research ( Site 0566), Escondido, California
  - Fresenius Kidney Care Newhope Fountain Valley ( Site 0617), Fountain Valley, California
  - DaVita Glendale Heights ( Site 0604), Glendale, California
  - DaVita West Glendale Dialysis ( Site 0579), Glendale, California
  - DaVita North Glendale ( Site 0552), Glendale, California
  - California Institute of Renal Research - La Mesa ( Site 0682), La Mesa, California
  - La Puente Dialysis Center ( Site 0610), La Puente, California
  - Academic Medical Research Institute ( Site 0533), Los Angeles, California
  - DaVita Kidney Center - East LA Plaza Dialysis ( Site 0548), Los Angeles, California
  - DaVita Crescent Heights Dialysis Center ( Site 0574), Los Angeles, California
  - North America Research Institute ( Site 0587), Lynwood, California
  - North America Research Institute ( Site 0612), Lynwood, California
  - Valley Renal Medical Group Research-Clinical Research ( Site 0651), Northridge, California
  - California Institute of Renal Research - Kearny Mesa ( Site 0678), San Diego, California
  - North America Research Institute ( Site 0611), San Dimas, California
  - DaVita Van Nuys Dialysis ( Site 0538), Van Nuys, California
  - Desert Cities Diaylsis-Clinical Research ( Site 0615), Victorville, California
  - DaVita Clinical Research - Hartford ( Site 0507), Hartford, Connecticut
  - DaVita Clinical Research - Middlebury ( Site 0511), Middlebury, Connecticut
  - Research Physicians Network Alliance ( Site 0563), Boca Raton, Florida
  - Horizon Research Group ( Site 0578), Coral Gables, Florida
  - Horizon Research Group ( Site 0581), Coral Gables, Florida
  - Elixia at Florida Kidney Physicians - Southeast ( Site 0602), Fort Lauderdale, Florida
  - South Florida Research Institute ( Site 0656), Fort Lauderdale, Florida
  - Elixia Clinical Research Collaborative (CRC) - Southeast Florida ( Site 0728), Hollywood, Florida
  - Pines Clinical Research ( Site 0605), Hollywood, Florida
  - Floridian Clinical Research, LLC ( Site 0684), Miami Lakes, Florida
  - Omega Research Orlando ( Site 0645), Orlando, Florida
  - Genesis Clinical Research, LLC ( Site 0585), Tampa, Florida
  - Genesis Clinical Research, LLC ( Site 0594), Tampa, Florida
  - Genesis Clinical Research, LLC ( Site 0680), Tampa, Florida
  - DaVita Clinical Research - Columbus ( Site 0532), Columbus, Georgia
  - Renal Physicians of Georgia ( Site 0577), Macon, Georgia
  - DaVita East Georgia Dialysis Unit ( Site 0536), Statesboro, Georgia
  - University of Chicago Medical Center-Medicine - Section of Nephrology ( Site 0595), Chicago, Illinois
  - Nephrology Specialists - Merrillville ( Site 0537), Merrillville, Indiana
  - Nephrology Specialists - Michigan City ( Site 0541), Michigan City, Indiana
  - Capital Nephrology ( Site 0596), Greenbelt, Maryland
  - Henry Ford Hospital-Nephrology and Hypertension ( Site 0694), Detroit, Michigan
  - St. Clair Nephrology Research - Roseville ( Site 0597), Roseville, Michigan
  - DaVita Clinical Research ( Site 0502), Minneapolis, Minnesota
  - Fresenius Kidney Care Brookhaven ( Site 0693), Brookhaven, Mississippi
  - Clinical Research Consultants, LLC ( Site 0542), Kansas City, Missouri
  - Somnos Clinical Research ( Site 0669), Lincoln, Nebraska
  - DaVita Five Star Dialysis Center ( Site 0509), Las Vegas, Nevada
  - Renal Medicine Associates ( Site 0690), Albuquerque, New Mexico
  - Capital District Renal Physicians ( Site 0633), Albany, New York
  - Ridgewood Dialysis Center ( Site 0725), Ridgewood, New York
  - Albert Einstein College of Medicine-Department of Medicine-Nephrology Einstein ( Site 0628), The Bronx, New York
  - DaVita Clinical Researh ( Site 0501), The Bronx, New York
  - Fresenius Kidney Care - Charlotte ( Site 0686), Charlotte, North Carolina
  - Durham Nephrology Associates ( Site 0655), Durham, North Carolina
  - East Carolina University-Department of Nephrology & Hypertension ( Site 0663), Greenville, North Carolina
  - Kidney and Hypertension Center ( Site 0571), Roseburg, Oregon
  - Northeast Clinical Research Center ( Site 0653), Bethlehem, Pennsylvania
  - Elixia at Clinical Renal Associates ( Site 0677), Upland, Pennsylvania
  - South Carolina Nephrology & Hypertension Center-Research ( Site 0672), Orangeburg, South Carolina
  - Knoxville Kidney Center ( Site 0689), Knoxville, Tennessee
  - Renal Disease Research Institute ( Site 0621), Dallas, Texas
  - DaVita Clinical Research - El Paso ( Site 0505), El Paso, Texas
  - DaVita Clinical Research - Houston ( Site 0508), Houston, Texas
  - Clinical Research Strategies ( Site 0625), Houston, Texas
  - Southwest Houston Research ( Site 0649), Houston, Texas
  - Texas Institute for Kidney and Endocrine Disorders ( Site 0626), Lufkin, Texas
  - Gamma Medical Research ( Site 0688), McAllen, Texas
  - DaVita Clinical Research - Norfolk ( Site 0513), Norfolk, Virginia
  - DaVita Clinical Research - Milwaukee ( Site 0512), Wauwatosa, Wisconsin
- Argentina (7):
  - FME Mansilla ( Site 0007), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fresenius Medical Care - Moron ( Site 0008), Morón, Buenos Aires
  - Fresenius Medical Care - San Fernando ( Site 0013), San Fernando, Buenos Aires
  - CEREHA ( Site 0004), Sarandí, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC) ( Site 0010), Buenos Aires, Buenos Aires F.D.
  - Fresenius Medical Care Ciudad Evita ( Site 0006), Buenos Aires
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares ( Site 0001), Santa Fe
- Western Health-Sunshine & Footscray Hospitals-Renal Services ( Site 0054), St Albans, Victoria, Australia
- Brazil (3):
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto-Centro Integrado de Pesquisa ( Site, São José do Rio Preto, São Paulo
  - Fresenius Clinical Trials Perdizes ( Site 0101), São Paulo, São Paulo
  - Hospital do Rim e Hipertensão ( Site 0106), São Paulo
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment - "Dr. Cherven Bryag"-Department of dialysis treatment (, Cherven Bryag, Lovech
  - MHAT Dobrich-Department for dialysis treatment ( Site 0161), Dobrich
  - First Dialysis Services Bulgaria ( Site 0158), Montana
  - UMBAL Plovdiv AD-Deparment of Hemodialysis ( Site 0162), Plovdiv
  - Hemomed ( Site 0159), Sofia
- Canada (2):
  - University Of Alberta Hospital ( Site 1001), Edmonton, Alberta
  - Toronto General Hospital ( Site 1002), Toronto, Ontario
- Czechia (3):
  - Fresenius Medical Care - Dialyzační středisko ( Site 0254), Prague, Praha 4
  - Dialýza ( Site 0256), Beroun
  - Fresenius Medical Care ( Site 0253), Pardubice
- DaVita Clinical Research Germany GmbH ( Site 0901), Düsseldorf, North Rhine-Westphalia, Germany
- Greece (3):
  - ATTIKON GENERAL UNIVERSITY HOSPITAL-2nd Dep. of Int. Medicine. Research Unit & Diabetes Center ( Sit, Chaïdári, Attica
  - Ippokrateio General Hospital of Thessaloniki ( Site 1053), Thessaloniki, Central Macedonia
  - G. Papanikolaou General Hospital-Nephrology Department ( Site 1052), Thessaloniki
- Italy (3):
  - P.O. San Carlo Borromeo- ASST SANTI PAOLO E CARLO ( Site 0954), Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0953), Milan
  - Fondazione Salvatore Maugeri clinica del lavoro ( Site 0955), Pavia
- Portugal (5):
  - Fresenius Medical Care - NephroCare Covilha ( Site 0852), Covilha, Castelo Branco District
  - Fresenius Medical Care - Nephrocare Portimao ( Site 0855), Portimão, Faro District
  - Fresenius Medical Care - NephroCare Amadora ( Site 0851), Amadora, Lisbon District
  - Fresenius Medical Care - NephroCare Almada ( Site 0854), Corroios, Lisbon District
  - Dyalisis Center - Clinic NephroCare Lumiar -Fresenius ( Site 0853), Lisbon, Lisbon District
- Fresenius Medical Care Humacao ( Site 0354), Humacao, Puerto Rico
- Romania (4):
  - Fresenius Nephrocare - Brașov ( Site 0409), Brașov, Brăila County
  - Fresenius Nephrocare - Bucharest ( Site 0408), Bucharest, București
  - Fresenius Nephrocare - Cluj-Napoca ( Site 0410), Cluj-Napoca, Cluj
  - Fresenius Nephrocare - Iași ( Site 0406), Iași, Iaşi
- Russia (2):
  - Unipharm LLC ( Site 0804), Krasnogorsk, Moscow Oblast
  - Limited Liability Company -Nefroline-Novosibirsk ( Site 0810), Novosibirsk, Novosibirsk Oblast
- Sweden (3):
  - Skånes Universitetssjukhus Malmö ( Site 0454), Malmo, Skåne County
  - Karolinska Universitetssjukhuset Huddinge-ME Njurmedicin ( Site 0451), Stockholm, Stockholm County
  - Akademiska sjukhuset-Njurmottagningen ( Site 0453), Uppsala, Uppsala County

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26294&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant with trial "Status Not Recorded" was discontinued from trial participation due to site termination of sponsor, but discontinuation form was not completed in the electronic data capture (EDC) in time by the terminated site.
Period: Overall Study
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo
Started | 171 | 167 | 168
Treated | 170 | 164 | 168
Completed | 105 | 113 | 113
Not Completed | 66 | 54 | 55
Not completed — Death | 47 | 42 | 39
Not completed — Withdrawal by Parent/Guardian | 1 | 0 | 0
Not completed — Site Terminated By Sponsor | 3 | 0 | 2
Not completed — Withdrawal by Subject | 13 | 8 | 10
Not completed — Lost to Follow-up | 2 | 4 | 3
Not completed — Status Not Recorded | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo | Total
Number analyzed (Participants) | 171 | 167 | 168 | 506
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (13.5) | 58.8 (12.8) | 60.5 (14.8) | 60.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 81 | 83 | 261
  Male | 74 | 86 | 85 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 67 | 65 | 209
  Not Hispanic or Latino | 91 | 98 | 100 | 289
  Unknown or Not Reported | 3 | 2 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 4
  Asian | 6 | 6 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 63 | 73 | 67 | 203
  White | 99 | 86 | 94 | 279
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region [Count of Participants; unit: Participants] — Participants were classified based on their geographic region as being either United States (US) or non-US.
  Participants
    US | 118 | 117 | 118 | 353
    non-US | 53 | 50 | 50 | 153
Previous Thrombosis of Active Arteriovenous Graft (AVG) [Count of Participants; unit: Participants] — Participants were classified based on having previous thrombosis of active AVG, with 'Yes' as having previous thrombosis of active AVG and 'No' as not having previous thrombosis of active AVG.
  Participants
    Yes | 38 | 35 | 40 | 113
    No | 133 | 132 | 128 | 393
Regular Aspirin Use up to 150 mg Daily at Baseline [Count of Participants; unit: Participants] — Participants were classified based on regular aspirin use up to 150 mg daily at baseline, with 'Yes' as regular use of aspirin up to 150 mg daily at baseline and 'No' as not having regular use of aspirin up to 150 mg daily at baseline.
  Participants
    Yes | 72 | 69 | 67 | 208
    No | 99 | 98 | 101 | 298

OUTCOME MEASURES:

1. Primary Outcome: Time to First Arteriovenous Graft (AVG) Thrombosis Event
Description: An AVG thrombosis event is defined as the sudden occlusion of the participant's AVG requiring thrombectomy/thrombolysis, or clinical evidence of thrombosis with surgical, radiological or pathological conformation of an AVG thrombosis. A blinded independent clinical adjudication committee (CAC) adjudicated AVG thrombosis events. A time-to-event methodology was used to evaluate the results. The incidence rate is presented.
Time Frame: From date of randomization until the date of first occurrence of an AVG thrombosis event, assessed up to approximately 37 months
Population: The analysis population consisted of all randomized participants, excluding three participants with arteriovenous fistula (AVF) rather than an AVG at randomization.
Measure: Number; unit: events per 100 person-years
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo
Number analyzed (Participants) | 171 | 165 | 167
events per 100 person-years | 23.80 | 22.98 | 30.17
Statistical Analysis 1: Comparison: MK-2060 20 mg vs Placebo; Test type: Superiority; p = 0.470, Log Rank — From log-rank test stratified by region (US, Non-US), previous thrombosis of active AVG (yes, no) and regular aspirin use up to 150 mg daily at baseline (yes, no); Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.60 to 1.26] — HR based on stratified Cox model with Efron's method of tie handling and with a single treatment covariate, controlling for stratification factors of region, previous thrombosis of active AVG and regular aspirin use up to 150 mg daily at baseline
Statistical Analysis 2: Comparison: MK-2060 6 mg vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.57 to 1.19] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time to Each AVG Thrombosis Event (First and Recurrent)
Description: An AVG thrombosis event is defined as the sudden occlusion of the participant's AVG requiring thrombectomy/thrombolysis, or clinical evidence of thrombosis with surgical, radiological or pathological conformation of an AVG thrombosis. A blinded independent CAC adjudicated AVG thrombosis events. A time-to-event methodology was used to evaluate the results. The incidence rate is presented.
Time Frame: Up to approximately 37 months
Population: The analysis population consisted of all randomized participants, excluding three participants with AVF rather than an AVG at randomization.
Measure: Number; unit: events per 100 person-years
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo
Number analyzed (Participants) | 171 | 165 | 167
events per 100 person-years | 38.95 | 37.85 | 42.97
Statistical Analysis 1: Comparison: MK-2060 20 mg vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.68 to 1.21] — HR based on Andersen-Gill model with stratification factors of region, previous thrombosis of active AVG, and regular aspirin use up to 150 mg daily at baseline as fixed effect
Statistical Analysis 2: Comparison: MK-2060 6 mg vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.70 to 1.23] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with one or more AEs is presented.
Time Frame: Up to approximately 40 months
Population: The analysis population consisted of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo
Number analyzed (Participants) | 170 | 164 | 168
Participants | 161 | 143 | 155

4. Secondary Outcome: Time to First Event of International Society on Thrombosis (ISTH) Major Bleeding Event or a Clinically Relevant Non-Major Bleeding Event
Description: Major bleeding events were defined as a having symptomatic presentation and including ≥1 of the following criteria: 1) Fatal bleeding 2) Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial, intramuscular with compartment syndrome 3) Bleeding causing decrease in hematocrit level of 20 g/L or more or leading to transfusion of ≥2 units of whole blood or red cells. Clinically relevant non-major bleeding events were defined as signs or symptoms of hemorrhage that do not meet criteria for major bleeding events but meet ≥1 of the following criteria: 1) Requiring medical intervention by healthcare professional 2) Leading to hospitalization or increased level of care 3) Prompting face-to-face evaluation by healthcare professional. A time-to-event methodology was used. The incidence rate is presented.
Time Frame: From date of first dose of study intervention until the first ISTH major bleeding event or a clinically relevant non-major bleeding event. assessed up to approximately 40 months
Population: The analysis population consisted of all randomized participants who received at least one dose of study intervention.
Measure: Number; unit: events per 100 person-years
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo
Number analyzed (Participants) | 170 | 164 | 168
events per 100 person-years | 24.73 | 18.05 | 14.04
Statistical Analysis 1: Comparison: MK-2060 20 mg vs Placebo; Test type: Other; p = 0.022, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.68, 95% CI 2-sided [1.07 to 2.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-2060 6 mg vs Placebo; Test type: Other; p = 0.311, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.800 to 2.00] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants Who Discontinue Study Intervention Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study intervention due to an AE is presented.
Time Frame: Up to approximately 37 months
Population: The analysis population consisted of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo
Number analyzed (Participants) | 170 | 164 | 168
Participants | 47 | 32 | 46

ADVERSE EVENTS:
Time Frame: Up to approximately 40 months
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) include all randomized participants who received ≥1 dose of study intervention.
Arm/Group | MK-2060 20 mg | MK-2060 6 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 50/171 | 43/167 | 41/168
Serious Adverse Events (participants affected / at risk) | 110/170 | 95/164 | 112/168
Other Adverse Events (participants affected / at risk) | 111/170 | 106/164 | 109/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2060 20 mg (N=170) | MK-2060 6 mg (N=164) | Placebo (N=168)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 2 (2) | 2 (3)
Acute myocardial infarction (Cardiac disorders) | 9 (10) | 6 (7) | 8 (8)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (4) | 5 (6)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (5) | 3 (3) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 10 (12) | 1 (2) | 5 (5)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart failure with preserved ejection fraction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (5) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Stomatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Accidental death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3)
Catheter site haemorrhage (General disorders) | 1 (1) | 2 (2) | 1 (1)
Chest pain (General disorders) | 3 (3) | 9 (11) | 2 (2)
Death (General disorders) | 4 (4) | 5 (5) | 5 (5)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 1 (1)
Gait inability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 1 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 6 (7) | 1 (1) | 2 (2)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial translocation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 7 (7) | 3 (3) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 4 (4) | 3 (4)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 4 (4) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2) | 6 (8) | 6 (7)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (13) | 9 (10) | 13 (14)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Polyomavirus-associated nephropathy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 4 (7) | 11 (12)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 4 (4) | 5 (5)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular access site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular graft infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft site complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 4 (4)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 13 (15) | 19 (24) | 19 (22)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Post procedural urine leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 (1) | 2 (4) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access site ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Coma scale abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (3) | 0 (0) | 3 (3)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (8) | 6 (6) | 12 (16)
Hypervolaemia (Metabolism and nutrition disorders) | 8 (13) | 9 (10) | 11 (16)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (4) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 3 (3) | 3 (3)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (9) | 5 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (17)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (3)
Renal transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 3 (3)
Therapy cessation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dialysis hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 2 (2) | 3 (3) | 3 (3)
Hypertensive urgency (Vascular disorders) | 0 (0) | 2 (3) | 3 (3)
Hypotension (Vascular disorders) | 5 (5) | 1 (1) | 3 (3)
Hypotensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Subclavian vein stenosis (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Venous occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2060 20 mg (N=170) | MK-2060 6 mg (N=164) | Placebo (N=168)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 2 (4) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 11 (12) | 11 (13) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 11 (17) | 20 (26) | 9 (11)
Nausea (Gastrointestinal disorders) | 9 (12) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 9 (9) | 6 (7) | 10 (11)
Chest pain (General disorders) | 10 (12) | 8 (8) | 10 (11)
Puncture site haemorrhage (General disorders) | 5 (12) | 9 (13) | 2 (5)
COVID-19 (Infections and infestations) | 13 (14) | 10 (10) | 18 (18)
Urinary tract infection (Infections and infestations) | 10 (12) | 7 (12) | 8 (11)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 9 (24) | 16 (29) | 7 (8)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 22 (31) | 23 (51) | 23 (39)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 29 (54) | 35 (66) | 43 (86)
Fall (Injury, poisoning and procedural complications) | 15 (15) | 11 (11) | 9 (18)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (10) | 10 (10) | 11 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (7) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (10) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (15) | 6 (6) | 9 (9)
Dizziness (Nervous system disorders) | 8 (17) | 3 (4) | 10 (10)
Headache (Nervous system disorders) | 9 (11) | 10 (13) | 14 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (10) | 16 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (17) | 6 (8) | 4 (4)
Hypertension (Vascular disorders) | 17 (20) | 9 (9) | 10 (21)
Hypotension (Vascular disorders) | 12 (12) | 7 (10) | 15 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT05027074/Prot_SAP_000.pdf